CLINICAL TRIAL: NCT05808374
Title: Phase I Clinical Study to Evaluate the Safety, Tolerance and Pharmacokinetic Characteristics of Single Administration of HRS-5635 Injection in Chinese Healthy Subjects and the Safety, Tolerance, Pharmacokinetics and Antiviral Effect of Multiple Administration in Patients With Chronic Hepatitis B
Brief Title: Clinical Study to Evaluate the Safety, Tolerance and Pharmacokinetic Characteristics of Single Administration of HRS-5635 Injection in Chinese Healthy Subjects and the Safety, Tolerance, Pharmacokinetics and Antiviral Effect of Multiple Administration in Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HRS-5635-101
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Single Dose Incremental (SAD) Trial - Healthy Persons：HRS-5635 vs. Placebo
  Interventions: Drug: HRS-5635; Drug: Placebo
- Part 2a (Experimental): Multiple Dose Increase (MAD) Study - Patients Receiving Consolidation Therapy：HRS-5635 vs. Placebo
  Interventions: Drug: HRS-5635; Drug: Placebo
- Part 2b (Experimental): Patients not receiving consolidation treatment：HRS-5635 vs. Placebo
  Interventions: Drug: HRS-5635; Drug: Placebo

INTERVENTIONS:
Drug: HRS-5635 — 50mg HRS-5635；100mg HRS-5635；200mg HRS-5635；400mg HRS-5635；600mg HRS-5635；800mg HRS-5635
  Arms: Part 1
Drug: HRS-5635 — 100mg HRS-5635，Q4W；200mg HRS-5635 ，Q4W；400mg HRS-5635，Q4W；200mg HRS-5635, Q2W
  Arms: Part 2a
Drug: HRS-5635 — 200mg HRS-5635，Q4W
  Arms: Part 2b
Drug: Placebo — Placebo

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS-5635 in healthy adults and chronic hepatitis B. To explore the reasonable dosage of HRS-5635.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the specific process of the test, voluntarily participate in the test, and sign the informed consent form in writing（In healthy people and chronic hepatitis B）.
2. Age 18-55 (including boundary value) （In healthy people）; Age 18-65 (including boundary value) （In chronic hepatitis B）.
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) 18~28 kg/m2 (including boundary value) （In healthy people）.
4. Normal or abnormal vital signs, physical examination, laboratory examination, chest radiograph, etc. have no clinical significance（In healthy people）.
5. Subjects (including partners) are willing to voluntarily take effective contraceptive measures within 6 months after screening and the last study drug administration（In healthy people）.

Exclusion Criteria:

1. Those suffering from any clinical serious disease such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormality, or any other disease that can interfere with the test results（In healthy people）.
2. Previous history of malignant tumor（In healthy people）.
3. Those who have digestive system disease or serious digestive system disease at present or in the near future (within one month), and the researcher believes that it may affect drug absorption or have safety risk（In healthy people）.
4. Those who have serious infection, serious injury or major surgery within 3 months before administration; Those who plan to undergo surgery during the trial and within two weeks after the end of the trial（In healthy people）.
5. Serious cardiovascular and cerebrovascular diseases with clinical significance and unstable or uncontrolled conditions, including but not limited to myocardial infarction, unstable angina pectoris, heart failure, and moderate stroke（（In chronic hepatitis B））.
6. Clinically significant liver diseases caused by other causes (such as alcoholic liver disease, nonalcoholic steatohepatitis, drug-induced liver injury, alcoholic hepatitis, etc.); （In chronic hepatitis B）.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events In Part 1 | 85 days
  A summary of adverse events, including Serious Adverse Events(SAEs)
Number of Adverse Events In Part 2 | 169 days
  A summary of adverse events, including Serious Adverse Events(SAEs)

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of single dose | 8 days
Peak Plasma Concentration (Cmax) of Multiple ascending dose | 64 days
Time to the peak plasma concentration (Tmax) of single dose | 8 days
Time to the peak plasma concentration (Tmax) of Multiple ascending dose | 64 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China University of Science and Technology, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided